CLINICAL TRIAL: NCT05725304
Title: National Health Research Institutes,Taiwan
Brief Title: The Registry of Genetic Expression of Taiwan Urologic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T1822
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Urologic Cancer
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — more than 30% of tumor compartments tissue. RCC arms (N=200): ccRCC (N=100) and nccRCC (N=100) or UC urinary tract (N=300). The study aims to obtain cancer tissues that originated from bladder (N=100), ureter (N=100), and renal pelvis (N=100).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- kidney cancer: RCC arms: Retrospective studies for ccRCC (N=100) and nccRCC (N=100). The studies aim to obtain clinical information to correlate with genetic characterization of RCCs of all types.
- urothelial cancer: UC arm: This is a prospective study for UC originated from the translational epithelium in the urinary tract (N=300). The study aims to obtain cancer tissues that originated from bladder (N=100), ureter (N=100), and renal pelvis (N=100).

SUMMARY:
This project is a nationwide precision medicine program for urothelial carcinoma and renal cell carcinoma.

DETAILED DESCRIPTION:
This project providing free and immediate next-generation gene sequencing testing for patients with urothelial and renal cell carcinomas that have is diagnosed or that have previously received systemic therapy. The goal of this project is to assist participating institutions in integrating next-generation sequencing results and building a real-time data storage and sharing platform, as well as establishing a tumor molecular biological atlas of Taiwanese patients with urothelial carcinoma and renal cell carcinoma. The data will be linked with clinical prognosis to facilitate the rapid screening of patients for effective potential therapeutic drugs and clinical trials, which is anticipated to prolong the survival rate of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20 and above. (Age >= 18 years old from January 1, 2023).
2. Pathological reports showed renal cell carinoma or urothelial carcinoma.
3. muscle-invasive bladder cancer or positive of N/M grade, UTUC of T2 at least or positive of N/M grade, or stage III/IV RCC
4. Willingness to provide the residual biopsy/operative tumor samples for study.
5. Life expectancy more than 3 months.
6. Patients fully understand the protocol with the willingness to have regular follow-up.

Exclusion Criteria:

1. Inability to cooperate by providing a complete medical history.
2. Ineligible tumor tissue samples for next-generation sequencing of genetic testing.
3. Undesirable compliance.
4. Having a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: urothelial carcinoma and renal cell carcinoma
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2029-10-29 (Estimated); Study Completion 2029-10-29 (Estimated)

PRIMARY OUTCOMES:
Development of an integrated database of genetic background | From date of registration to 30 Sep 2029
  Development of an integrated database of genetic background from populations, underlying status, clinical information, and therapeutic outcomes in carcinogen-related advanced urologic tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Lung Cha, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Yu wei-lan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will be linked with clinical prognosis to facilitate the rapid screening of patients for effective potential therapeutic drugs and clinical trials, which is anticipated to prolong the survival rate of patients.